CLINICAL TRIAL: NCT05693077
Title: Establishing Colonisation With Non-toxigenic Clostridioides Difficile in Healthy Volunteers
Brief Title: Clostridioides Difficile Colonisation
Acronym: CloDiCo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof. dr., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CloDiCo
Record Dates: First submitted 2022-12-21; First posted 2023-01-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Clostridioides Difficile Infection
Keywords: Colonization
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: The trial consists of two or, if necessary, three consecutive intervention phases with each three parallel intervention arms. The first phase consists 24 volunteers, the second phase of 23 or 26 volunteers, and the optional third phase of another 23 volunteers. The volunteers will be divided over three intervention arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is double-blind, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group A (phase 1) (N=10) (Experimental): 5 doses of 10E4 NTCD spores on day 0-4.
  Interventions: Biological: 10E4 NTCD spores
- Group B (phase 1) (N=10) (Experimental): 5 doses of 10E7 NTCD spores on day 0-4.
  Interventions: Biological: 10E7 NTCD spores
- Group C (phase 1) (N=4) (Placebo Comparator): 5 doses of placebo on day 0-4.
  Interventions: Other: placebo
- Group D (phase 2) (N=10) (Experimental): Based upon the colonisation results of phase 1, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all three groups in phase 2:
  * Option 1: 3 doses of 10E4 NTCD spores on day 0-2.
  * Option 2: 3 doses of 10E7 NTCD spores on day 0-2.
  * Option 3: 1 day of vancomycin on day -7, followed by 5 doses of 10E4 NTCD spores on day 0-4.
  Interventions: Biological: 10E4 NTCD spores; Biological: 10E7 NTCD spores; Drug: Vancomycin Oral Capsule
- Group E (phase 2) (N=10) (Experimental): Based upon the colonisation results of phase 1, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all three groups in phase 2:
  * Option 1: 1 dose of 10E4 NTCD spores on day 0, and 2 doses of placebo on day 1-2.
  * Option 2: 1 dose of 10E7 NTCD spores on day 0, and 2 doses of placebo on day 1-2.
  * Option 3: 1 day vancomycin on day -7 followed by 5 doses of 10E7 NTCD spores on day 0-4.
  Interventions: Biological: 10E4 NTCD spores; Biological: 10E7 NTCD spores; Other: placebo; Drug: Vancomycin Oral Capsule
- Group F (phase 2) (N=3 or 6) (Placebo Comparator): Based upon the colonisation results of phase 1, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all of the groups:
  * Option 1 (N=6): 3 doses of placebo on day 0-2.
  * Option 2 (N=6): 3 doses of placebo on day 0-2.
  * Option 3 (N=3): 1 day vancomycin on day -7, followed by 5 doses of placebo on day 0-4.
  Interventions: Other: placebo; Drug: Vancomycin Oral Capsule
- Group G (phase 3) (N=10) (Experimental): Escalation to the third phase will only be done if option 3 is selected in phase 2. Based upon the colonisation results of phase 2, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all of the groups in phase 3:
  * Option 1: 1 day vancomycin on day -7, followed by 3 doses of 10E4 NTCD spores on day 0-2.
  * Option 2: 1 day vancomycin on day -7, followed by 3 doses of 10E7 NTCD spores on day 0-2.
  * Option 3: 5 days of vancomycin on day -11 until day -7, followed by 5 doses of 10E4 NTCD spores on day 0-4.
  Interventions: Biological: 10E4 NTCD spores; Biological: 10E7 NTCD spores; Drug: Vancomycin Oral Capsule
- Group H (phase 3) (N=10) (Experimental): Escalation to the third phase will only be done if option 3 is selected in phase 2. Based upon the colonisation results of phase 2, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all of the groups in phase 3:
  * Option 1: 1 day of vancomycin on day -7, followed by 1 dose of 10E4 NTCD spores on day 0, and 2 doses of placebo on day 1-2.
  * Option 2: 1 day of vancomycin on day -7, followed by 1 dose of 10E7 NTCD spores on day 0 and 2 doses of placebo on day 1-2.
  * Option 3: 5 days of vancomycin on day -11 until day -7, followed by 5 doses of 10E7 NTCD spores on day 0-4.
  Interventions: Biological: 10E4 NTCD spores; Biological: 10E7 NTCD spores; Other: placebo; Drug: Vancomycin Oral Capsule
- Group I (phase 3) (N=3) (Placebo Comparator): Escalation to the third phase will only be done if option 3 is selected in phase 2. Based upon the colonisation results of phase 2, there are three dosing options for this group, one of the three options will be chosen, the chosen option number will be congruent for all of the groups in phase 3:
  * Option 1: 1 day of vancomycin on day -7, followed by 3 doses of placebo on day 0-2.
  * Option 2: 1 day of vancomycin on day -7, followed by 3 doses of placebo on day 0-2.
  * Option 3: 5 days of vancomycin on day -11 until day -7, followed by 5 doses of placebo on day 0-4.
  Interventions: Other: placebo; Drug: Vancomycin Oral Capsule

INTERVENTIONS:
Biological: 10E4 NTCD spores — in capsule for oral ingestion.
  Arms: Group A (phase 1) (N=10); Group D (phase 2) (N=10); Group E (phase 2) (N=10); Group G (phase 3) (N=10); Group H (phase 3) (N=10)
Biological: 10E7 NTCD spores — in capsule for oral ingestion.
  Arms: Group B (phase 1) (N=10); Group D (phase 2) (N=10); Group E (phase 2) (N=10); Group G (phase 3) (N=10); Group H (phase 3) (N=10)
Other: placebo — in capsule for oral ingestion.
  Arms: Group C (phase 1) (N=4); Group E (phase 2) (N=10); Group F (phase 2) (N=3 or 6); Group H (phase 3) (N=10); Group I (phase 3) (N=3)
Drug: Vancomycin Oral Capsule — 4 times a day 250mg
  Arms: Group D (phase 2) (N=10); Group E (phase 2) (N=10); Group F (phase 2) (N=3 or 6); Group G (phase 3) (N=10); Group H (phase 3) (N=10); Group I (phase 3) (N=3)

SUMMARY:
This study will investigate experimental colonisation with non-toxigenic C.difficile (NTCD) in healthy volunteers. Main outcomes will be safety, tolerability, dose needed to obtain colonisation with NTCD to ultimately determine host microbiota factors associated with susceptibility to colonisation.

DETAILED DESCRIPTION:
This will be an adaptive dose design, randomized double-blind controlled clinical trial investigating oral exposure to NTCD spores in healthy volunteers. The trial will consist of two or, if necessary, three different consecutive intervention phases. The second and third phase are dependent on results of the preliminary phases. In every phase one cohort volunteers will be randomized to different dose levels of NTCD spores or placebo.

50 to 70 healthy volunteers will be included, of which in total 10 volunteers will be exposed to placebo.

The first phase will consist of 24 volunteers, randomized in three groups: group A (N=10) will receive 5 doses of 10E4 NTCD spores, group B (N=10) will receive 5 doses of 10E7 NTCD spores and group C (N=4) will receive 5 doses of placebo.

Depending on the outcome of phase 1, the dose given in phase 2 will either be reduced (if colonisation frequency in phase 1 is >60%), or the doses will be preceded by vancomycin pre-treatment (if the colonisation frequency in phase 1 is <60%) according to predefined criteria. There are three dosing options for phase 2: for the first two options (reduced doses of NTCD) 26 volunteers will be divided over 3 groups group D (N=10), group E (N=10) and the control group F (N=6), for the third option (vancomycin pre-treatment) 23 volunteers will be divided over 3 groups; group D (N=10), group E (N=10) and the control group F (N=3). For the dosing schedules of the three options op the second phase please refer to the section below 'Arms and Interventions'.

Escalation to the third phase will only be done if option 3 is selected in phase 2.Depending on the outcome of phase 2, the dose given in phase 3 will either be reduced (if colonisation frequency in phase 2 is >60%) or the vancomycin pre-treatment will be extended to five days (if the colonisation frequency in phase 2 is <60%) according to predefined criteria. 23 volunteers will be divided over 3 groups: group G (N=10), group H (N=10) and the control group I (N=3). For dosing schedules of the three options of the third phase please refer to the section below 'Arms and Interventions'.

All volunteers in all phases will visit the trial center on the days of spores or placebo ingestion (and if needed also on the first day of vancomycin ingestion), with collection of feces for C.difficile and microbiota analysis before ingestion. During the four follow-up weeks volunteers will visit the trial center three times a week for fecal sample collection (for Cdiff and microbiota analysis), with weekly follow-up visit for AE collection and 2 times a safety blood tests. After three months there will be a final follow-up visit for AEs and fecal sample collection. Should a volunteer still be positive for C.difficile at the three month timepoint, the volunteer is asked to return for follow-up every one to two months for fecal sample collection until the sample is negative for C.difficile, up till a maximum of one year after the start of the trial. Because colonisation with NTCD is very common in the general population, NTCD colonisation will not be terminated with antibiotics. Antibiotic rescue treatment (or in case of persistent disturbances to the host microbiota, a fecal microbiota transplantation) for NTCD is available in case of unexpected adverse events.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and is able and willing to abide strictly thereby.
3. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
4. Subject has signed informed consent.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any physical or psychiatric illness or conditions that could threaten or compromise the health of the subject during the study, influence their ability to participate in the trial or interfere with the interpretation of the study results, as determined by the trial physician.
2. Use of antibiotics (or other microbiota influencing products) within one month prior to inclusion.
3. Known immunosuppressive condition, including infection with Human Immunodeficiency Virus (HIV), use of systemic corticosteroids or other immune modifying drugs (with exception of antihistamines and topical steroids).
4. Regular use (defined by more than once weekly) of proton-pump inhibitors or H2- blockers during one month prior to inclusion.
5. The use of strong P-glycoprotein-inhibitors (like Ciclosporin, Ketoconazole, Erythromycin, Clarithromycin, Verapamil and Amiodaron).
6. Known allergy to vancomycin, metronidazole or fidaxomicin.
7. Known allergy to glycerol.
8. Known immunodeficiency disorders.
9. Known gastro-intestinal disease including but not limited to inflammatory bowel diseases (Crohn's disease, Colitis Ulcerosa), recent gastro-intestinal surgery, constipation defined by bowel movements less than every second day.
10. Positive fecal PCR with Clostridiodes or SSYC (Salmonella, Shigella, Yersinia or Campylobacter spp.) at screening.
11. Any condition that would put household members at a greater risk for transmission e.g. no access or use of flush toilet, household members belonging to vulnerable populations such as persons who are immunocompromised, children younger than 2 years of age and elderly older than 70 years of age.
12. For women of child bearing potential: a positive urine pregnancy test before inclusion or lactating at screening / during the trial.
13. Being an employee or student of the Experimental bacteriology group or the controlled human infection center at LUMC.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of colonisation with non-toxigenic C.difficile | During the first month after ingestion of NTCD spores.
  Number and grade of related adverse events from day 1 to 28 after ingestion of NTCD spores.
To establish the effective protocol to obtain colonisation with non-toxigenic C. difficile in the majority of subjects. | During the first month after ingestion of NTCD spores.
  The number of volunteers successfully colonised with non-toxigenic C.difficile. Colonisation is defined as a positive PCR for C.difficile on stool or a positive culture for C.difficile on at least two timepoints between three days and two weeks after the last exposure day.

SECONDARY OUTCOMES:
To determine factors in the host microbiota associated with successful colonisation. | 3 months after ingestion of NTCD spores.
  Microbiota markers which are associated with successful C.difficile colonisation through microbiota analysis with 16S amplicon sequencing.

OTHER OUTCOMES:
Determine changes in the host microbiota following colonisation. | 3 months after ingestion of NTCD spores.
  Identification of changes in microbiota components following C.difficile colonisation through microbiota analysis with 16S amplicon sequencing.
Investigate C. difficile in-vivo evolution. | 3 months after ingestion of NTCD spores.
  Identification of genetic changes of C.difficile after passage through the human host through C.difficile PCR and culturing.

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No